CLINICAL TRIAL: NCT04560920
Title: Enhancing Geriatric Pain Care With Contextual Patient Generated Data Profiles
Brief Title: Enhancing Geriatric Pain Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 19-265
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Pain
Keywords: patient generated health data; geriatrics; pain; contextual data; patient centered care; adherence
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: During aim 3, participants will be randomized to experimental or control group. Both groups will contribute PGHD, but the availability of PGHD at the visit will be the basis on which groups are compared. Earlier aims are not randomized but total anticipated enrollment is listed below.
Who Masked: Participant
Masking Description: Participants will be informed that they are participating in a study of patient information and that this information will be discussed when available at the visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): This group will contribute PGHD and it will be available in the study visit.
  Interventions: Other: Availability of contextual PGHD at the visit
- Control (No Intervention): This group may contribute PGHD but if so, it will not be available during a study visit, it will be available to the provider in a subsequent visit.

INTERVENTIONS:
Other: Availability of contextual PGHD at the visit — Contextual PGD will be available in a display at the visit.
  Arms: Experimental

SUMMARY:
This project is focused on Veteran patients 65 and older with chronic pain. In this project, the investigators will understand the impact of a contextual patient generated health data (PGHD). Contextual PGHD are data about what is important to patients, information about the Veterans social and home contexts (for example, how the Veterans medications are stored and how much help they receive from others). In this study the investigators will talk with Veterans with chronic pain and the Veterans informal caregivers (family members or friends who help them) and find out about how they are coping with chronic pain and what information might be helpful to provide to the Veterans healthcare team. Then, the investigators will talk to clinicians about information that might be helpful to them. The investigators will collect contextual PGHD and use it to develop a computer application for collecting contextual PGHD and displaying it to patients and doctors in a visit. The investigators will also test the impact of having contextual PGHD in a visit on patient satisfaction with the Veterans care plan and how well they are able to follow the care plan.

DETAILED DESCRIPTION:
The investigators proposal addresses the use of patient generated health data (PGHD) - an innovative approach to deliver patient centered care to older Veterans that is characterized by attention to patient priorities, values, and goals. The investigators clinical focus is on chronic pain in older Veterans, which is widespread. PGHD broadly encompasses many sources and types of data. The investigators will categorize contextual PGHD into 3 core components 1) relational PGHD (patient-clinician relationship and patient individual differences such as pain catastrophizing) 2) whole person PGHD (what matters to the patient including patient preferences), and 3) behavioral PGHD (pain self-efficacy and patient actions related to health , pain management, functional status). The investigators study is mixed methods.

In aim 1 the investigators will: Prioritize content for contextual PGHD profile displays to support patient centered care for geriatric Veterans with chronic pain. The investigators will conduct focus groups or interviews with geriatric Veterans with chronic pain and the Veterans caregivers to explore Veterans' perspectives on the content of the PGHD profile displays and the Veterans attitudes toward them. The investigators will conduct focus groups with clinicians about desired content of the PGHD profile displays specific to pain management. The investigators will iteratively prioritize PGHD elements in accordance with pain care management needs of geriatric patients, incorporating results of a card sort exercise performed by clinicians.

In aim 2 the investigators will :Develop a prototype contextual PGHD profile display and evaluate its usability. The investigators will develop a prototype clinician-facing PGHD profile display containing PGHD elements and guides to interpretation/use for clinicians. The investigators will refine the PGHD profile display prototype with clinicians in user-centered design sessions. The investigators will broadly assess usability in a simulation study with primary care clinicians.

In aim 3 the investigators will: Examine the impact of contextual PGHD profile displays on patient adherence, pain function, satisfaction, and shared decision making in a randomized trial. The investigators will evaluate operationalization of the pain care plan and the shared decision making process in the visit by coding study visit recordings. The investigators will assess the impact of contextual PGHD by comparing patient adherence to pain care regimens, pain function, patient satisfaction, and shared decision making process for a sample of 150 geriatric patients with chronic pain in VA primary care clinics. The investigators will compare between-subjects visits that include access to contextual PGHD profile displays to visits without access.

The investigators primary hypothesis is that access to contextual PGHD profile displays during a clinical visit will result in better adherence to the pain care plan at 30 days, compared with no PGHD profile display.

Throughout the project the investigators will work with stakeholders in clinic settings and implementation of the electronic health record to ensure future implementation can be optimized.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians are eligible if they are a primary care clinician or PACT member
* including physicians, nurse practitioners, nurses, social workers, pharmacists, and psychologists for Veteran patients over age 65 diagnosed with chronic pain in primary care, geriatrics clinic, or a local or rural CBOC within the Salt Lake City catchment.

Eligible VHA patients will be age 65 and older with a diagnosis of chronic pain defined by ICD 10 codes. Veteran caregivers (including spouses, other relatives, or close friends involved in the daily life of the Veteran) will also be eligible for participation in this study. Vulnerable populations, women, and minorities are eligible to the extent that they are represented in the above described population or are a caregiver.

Exclusion Criteria:

- Veterans who need a legally authorized representative to consent.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 230 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Adherence to the Pain Care Plan | Between 2 years and 4.5 years after study start
  MOS General Adherence Scale-Participants rate adherence on a 1-5 scale with higher scores indicating better adherence

SECONDARY OUTCOMES:
Patient Satisfaction with the Visit | 1.5 years to 4 years after study start
  SHEP communication scale, 4 items used to assess satisfaction with visit communication
Shared Decision Making in the Visit | 1.5 years to 4 years after study start
  Participatory Decision making style questionnaire, used in Medical Outcomes Study and relates to satisfaction with care. Participants rate participation on a 1-5 scale with higher scores indicating higher participation
Shared Decision Making in the visit | 1.5 years to 4 years after study start
  OPTION coding, a standardized coding scheme to capture shared decision making in the visit.
Pain Function | Between 2 years and 4.5 years after study start
  West Haven Yale Multidimensional Pain Inventory (WHYMPI). WHYMPI Statements are rated on a 0-6 Likert scale with higher scores indicating higher intensity
Patient perspective of Shared Decision Making | Between 2 years and 4.5 years after study start
  OPACIC adapted for older adults from the Patient Assessment of Chronic Illness Scale. This measure includes 5 subscales, patient activation, deliver system design/decision support, goal setting and tailoring, and follow-up/coordination. OPACIC statements are rated on a 1-5 Likert scale with higher scores indicating higher intensity

CONTACTS AND LOCATIONS:
Overall Officials: Jorie Butler, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT04560920/ICF_000.pdf